CLINICAL TRIAL: NCT00861913
Title: Phase II Trial of Pazopanib (GW786034) in Pre-Treated and Untreated Metastatic Melanoma Patients
Brief Title: Pazopanib Hydrochloride in Treating Patients With Metastatic Melanoma That Cannot be Removed by Surgery
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-01163; NCI-2009-01163 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000637188; MAYO-MC0875; MC0875 (Other: Mayo Clinic); 8218 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2009-03-13; First posted 2009-03-16 (Estimated); Results first posted 2014-01-21 (Estimated); Last update posted 2018-10-16 (Actual); Status verified 2018-09

CONDITIONS: Recurrent Melanoma; Stage IV Cutaneous Melanoma AJCC v6 and v7
MeSH Terms: conditions — Melanoma | interventions — pazopanib

ARMS (1):
- Treatment (pazopanib hydrochloride) (Experimental): Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given orally
  Other Names: GW786034B; Votrient
Other: Pharmacological Study — Correlative studies

SUMMARY:
This phase II trial is studying the side effects of pazopanib hydrochloride and to see how well it works in treating patients with metastatic melanoma that cannot be removed by surgery. Pazopanib hydrochloride may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the anti-tumor activity and safety profile of single agent Pazopanib (pazopanib hydrochloride).

SECONDARY OBJECTIVES:

I. To assess the impact of Pazopanib on circulating levels of vascular endothelial growth factor (VEGF).

II. To examine the association between tumor response and B-Raf and N-Ras mutations.

III. To examine pre/post-treatment expression levels of VEGF, vascular endothelial growth factor receptor (VEGFR)-1, VEGFR-2, VEGFR-3, and Ki67.

IV. To correlate baseline and changes in p-ERK levels in the tumor with response.

V. To determine pazopanib steady-state trough plasma concentrations (Css,min) and the relationships between Css,min and the PD effects and toxicities of pazopanib.

VI. To examine the associations of common polymorphisms in CYP1A2, CYP2C8, UGT1A1, ABCB1, and ABCG2 with the PK and PD of pazopanib.

VII. To Assess Progression Free Survival. VIII. To Assess Overall Survival.

OUTLINE: This is a multicenter study.

Patients receive oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

Patients undergo tumor tissue biopsy at baseline and blood sample collection at baseline and on days 14, 28, and 42 for research studies. Tumor tissue samples are analyzed by DNA sequencing, ELISA, western blotting, and immunoperoxidase staining. Blood samples are analyzed for pharmacodynamics, pharmacokinetics, and pharmacogenetics by high-performance liquid chromatography with tandem mass spectrometry.

After completion of study treatment, patients are followed periodically for up to 5 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed unresectable malignant melanoma

  * Radiographic or clinical evidence of metastatic disease
* Measurable disease with ≥ 1 lesion whose longest diameter can be measured as ≥ 2.0 cm by CT or MRI scans or ≥ 1.0 cm by spiral CT scan

  * Disease that is measurable by physical examination only is not allowed
* No known intraluminal metastatic lesion(s) with suspected bleeding
* No brain metastases by MRI or CT scan
* ECOG performance status 0-2
* Life expectancy > 12 weeks
* WBC ≥ 3,000/μL
* Hemoglobin ≥ 9 g/dL
* Absolute neutrophil count ≥ 1,500/μL
* Platelets ≥ 100,000/μL
* Total bilirubin ≤ 1.5 times upper limit of normal (ULN)
* AST and ALT ≤ 2.5 times ULN
* Creatinine ≤ 1.5 times ULN
* Serum troponin normal
* Urine protein ≤ 1+ (≤ 30 mg/dL) on 2 consecutive dipstick or other urine assessments taken ≥ 1 week apart
* QTc interval < 480 msec
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No significant ECG abnormalities (e.g., frequent ventricular ectopy, evidence of ongoing myocardial ischemia)
* No serious nonhealing wound, ulcer, or bone fracture
* No history of abdominal fistula, gastrointestinal perforation, active diverticulitis, intra-abdominal abscess, or gastrointestinal tract bleeding within the past 28 days
* No history of myocardial infarction, cardiac arrhythmia within the past 6 months
* No NYHA class III-IV heart failure

  * Patients with a history of class II heart failure and who are asymptomatic on treatment may be eligible
* No history of bleeding disorder, including hemophilia, disseminated intravascular coagulation, or any other abnormality of coagulation potentially predisposing patients to bleeding
* No uncontrolled infection
* No evidence of active bleeding or bleeding diathesis
* No hemoptysis within 6 weeks of first dose of study drug
* No active peptic ulcer disease
* No inflammatory bowel disease
* No ulcerative colitis or other gastrointestinal conditions with increased risk of perforation
* No history of cerebrovascular accident, including transient ischemic attack, pulmonary embolism, or untreated deep venous thrombosis within the past 6 months

  * Patients with recent deep vein thrombosis who have been treated with therapeutic anticoagulating agents within the past 6 weeks are eligible
* No known endobronchial lesions or involvement of large pulmonary vessels by tumor
* No current active hepatic or biliary disease, except Gilbert syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease
* No uncontrolled hypertension (i.e., systolic blood pressure [BP] > 140 mm Hg and diastolic BP > 90 mm Hg)
* No condition that impairs ability to swallow and retain pazopanib hydrochloride (e.g., gastrointestinal tract disease resulting in an inability to take oral medication or a requirement for IV alimentation, prior surgical procedures affecting absorption, or active peptic ulcer disease)
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or other agents used in the study
* No uncontrolled intercurrent illness including, but not limited to, ongoing or active infection or psychiatric illness/social situations that would or might reasonably be expected to limit compliance with study requirements
* No admission for unstable angina, cardiac angioplasty, or stenting within the past 6 months
* More than 6 weeks since prior major surgery
* More than 4 weeks since prior and no concurrent radiotherapy
* At least 14 days or 5 half-lives and no concurrent CYP interactive medications
* No prior radiotherapy to ≥ 25% of bone marrow
* No prior therapy with a VEGFR tyrosine-kinase inhibitor
* No concurrent antiretroviral therapy for HIV-positive patients
* No concurrent medications or substances known to affect or with the potential to affect the activity or pharmacokinetics of pazopanib hydrochloride
* No concurrent chemotherapy
* No other concurrent investigational agents
* No other concurrent anticancer agents or therapies
* No concurrent medications that are associated with a risk of QTc prolongation and/or Torsades de Pointes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2009-04-03 (Actual); Primary Completion 2010-09-14 (Actual); Study Completion 2014-01-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy Weise, Principal Investigator — Mayo Clinic
Locations (4):
- United States (4):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: From April 2009 to July 2009, 13 participants were registered.
Pre-assignment Details: All participants were evaluable for all endpoints and toxicity.
Groups:
- Treatment (Pazopanib Hydrochloride): Patients receive 800 mg oral pazopanib hydrochloride once daily on days 1-28. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Treatment (Pazopanib Hydrochloride)
Started | 13
Completed | 13
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 13
Age, Continuous [Median (Full Range); unit: years] | 64 [24 to 86]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 10
Region of Enrollment [Number; unit: participants]
  United States | 13

OUTCOME MEASURES:

1. Primary Outcome: Tumor Response Rate
Description: Tumor response rate is defined as the number of eligible patients whose disease status meets the Response Evaluation Criteria In Solid Tumors (RECIST) criteria for compete response (CR) or partial response (PR) divided by the number of evaluable patients. A ninety percent confidence interval for the true response proportion will be calculated assuming that the number of confirmed tumor responses follows a binomial distribution and using the Duffy-Santner approach.
  Complete Response (CR): Disappearance of all target lesions.
  Partial Response (PR): At least a 30% decrease in the sum of the largest dimension (LD) of target lesions taking as reference the baseline sum LD.
Time Frame: Up to 5 years
Measure: Number (90% Confidence Interval); unit: percentage of patients
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 13
percentage of patients | 7.7 [0.39 to 31.6]

2. Primary Outcome: Toxicity
Description: Toxicity is defined as any grade 3 or higher adverse event as assessed using the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 3.0 and at least possibly related to treatment. The maximum grade for each type of toxicity will be recorded for each patient. We report the number of patients experiencing a grade 3 or higher adverse event at least possibly related to treatment.
Time Frame: Up to 5 years
Measure: Number; unit: participants
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 13
participants
  Grade 3 | 8
  Grade 4 or higher | 0

3. Secondary Outcome: Overall Survival
Description: Overall survival time is defined as the time from registration to the time of death due to any cause. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to death due to any cause, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 13
months | 13.6 [6.0 to 18.6]

4. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from registration to the time of progression or death, whichever occurs first. Estimated using the method of Kaplan-Meier.
Time Frame: From registration to documentation of disease progression, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 13
months | 3.9 [1.8 to 4.0]

5. Secondary Outcome: Duration of Response
Description: The date at which the objective status is first noted to be either a Complete Response (CR) or Partial Response (PR) to the date progression is documented, assessed up to 5 years.
Time Frame: From time of documented response to the date progression is documented, assessed up to 5 years.
Population: There was one response and therefore median duration of response was not analyzed.
Arm/Group | Treatment (Pazopanib Hydrochloride)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Arm/Group | Treatment (Pazopanib Hydrochloride)
Serious Adverse Events (participants affected / at risk) | 5/13
Other Adverse Events (participants affected / at risk) | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 1 (2)
Hypothyroidism (Endocrine disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Leukocyte count decreased (Investigations) | 2 (3)
Neutrophil count decreased (Investigations) | 1 (2)
Platelet count decreased (Investigations) | 2 (3)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pazopanib Hydrochloride) (N=13)
Hemoglobin decreased (Blood and lymphatic system disorders) | 7 (15)
Hypothyroidism (Endocrine disorders) | 3 (5)
Eye disorder (Eye disorders) | 1 (1)
Vision blurred (Eye disorders) | 2 (3)
Abdominal pain (Gastrointestinal disorders) | 1 (4)
Constipation (Gastrointestinal disorders) | 1 (3)
Diarrhea (Gastrointestinal disorders) | 8 (37)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 1 (1)
Intra-abdominal hemorrhage (Gastrointestinal disorders) | 1 (1)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Mucositis oral (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (16)
Oral hemorrhage (Gastrointestinal disorders) | 1 (1)
Oral pain (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (2)
Vomiting (Gastrointestinal disorders) | 4 (6)
Edema limbs (General disorders) | 1 (1)
Fatigue (General disorders) | 13 (48)
Fever (General disorders) | 2 (2)
Pain (General disorders) | 1 (1)
Gingival infection (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 2 (3)
Amylase increased (Investigations) | 1 (2)
Bilirubin increased (Investigations) | 1 (2)
Leukocyte count decreased (Investigations) | 5 (20)
Neutrophil count decreased (Investigations) | 4 (11)
Platelet count decreased (Investigations) | 4 (23)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 8 (11)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 2 (2)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (2)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Taste alteration (Nervous system disorders) | 5 (13)
Anxiety (Psychiatric disorders) | 1 (3)
Depression (Psychiatric disorders) | 1 (1)
Cystitis (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 2 (16)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (1)
Rash desquamating (Skin and subcutaneous tissue disorders) | 1 (4)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 3 (18)
Hemorrhage (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 4 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less